CLINICAL TRIAL: NCT05942417
Title: Effects of Echoguided Percutaneous Neuromodulation (EPNM) of the Common Peroneal Nerve and Neuromuscular Exercise in the Management of Chronic Ankle Instability (CAI): a Randomized Clinical Trial (RCT).
Brief Title: Echoguided Percutaneous Neuromodulation in the Management of Chronic Ankle Instability in Physically Active Subjects.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escoles Universitaries Gimbernat (Other)
Collaborators: Universidad Rey Juan Carlos (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023137
Record Dates: First submitted 2023-06-26; First posted 2023-07-12 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Transcutaneous Electric Nerve Stimulation; Ankle Injuries and Disorders : Chronic Ankle Instability; Exercise Therapy
Keywords: Ankle; exercise therapy; chronic ankle instability; echoguided percutaneous neuromodulation
MeSH Terms: conditions — Ankle Injuries | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistical analysis investigator will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromodulation Percutaneous echoguided plus exercise (Experimental): The experimental group will receive a EPNM in the common peroneal nerve of the affected ankle. . Three interventions will be carried out, in a dosage of 1 per week. Moreover, a 3-week of strength exercises will be carried out with two sessions per week. The strength program includes a protocol for the use of Theraband ® according to that described by Kaminsky et al. Moreover, the participants will have to do a balance exercises program.The EPNM will be applied prior to the exercise program session
  Interventions: Procedure: Echoguided percutaneous neuromodulation plus exercise
- Strength program (Active Comparator): The strength program includes a Theraband® use protocol as described by Kaminsky et al.
  The balance exercise program will consist of performing a series of closed kinetic chain exercises in a weight-bearing standing position that will progress from bilateral to unilateral depending on the acceptance of the load.
  Interventions: Procedure: Strength program

INTERVENTIONS:
Procedure: Echoguided percutaneous neuromodulation plus exercise — This group is taking the EPNM and the exercise program
  Arms: Neuromodulation Percutaneous echoguided plus exercise
Procedure: Strength program — This group is taking the exercise program
  Arms: Strength program

SUMMARY:
The lateral ankle complex sprain is the most prevalent musculoskeletal injury among the general population and athletes and is associated with long-term pain, disability, and high healthcare costs. One of the complications of a lateral ankle sprain is the development of chronic ankle instability (CAI). Conservative treatment is the initial therapeutic option for patients with CAI, however, the best strategies are not yet clear. Clinically, a new invasive technique has appeared, known as echoguided Percutaneous Neuromodulation (EPNM). To date there are no studies showing the efficacy of the technique in patients with CAI together with the combination of a neuromuscular exercise program.

Participants: Volunteers and adults, from the group of students of the Gimbernat University School with a history of ankle sprain and physically active who meet the inclusion criteria.

Study variables: Self-administered ankle function scales (Cumberland ankle instability tool: CAIT and foot and ankle ability:FAAM measure Scale), objective measurement of function in the lower limb (Test countermovement jump: CMJ and Side hop Test:SHT), measurement of isometric strength of the ankle musculature, measurement of dynamic balance (Test star excursion balance), range of motion measurement (Ankle Dorsiflexion) and pain measurement (Numeric pain rating scale: NPRS Scale).

Procedures: After carrying out the assessment, the participants will be randomized to participate in a neuromuscular exercise intervention (control group) or in a neuromuscular exercise intervention together with an application of EPNM in the common peroneal nerve (control group). experimental). The duration of the intervention in both cases will be 3 weeks, where in the control group there will be 2 sessions per week of exercise and in the experimental group 2 sessions per week of exercise plus an application of EPNM.

Objective and hypothesis: The main objective of the study will be to compare the short- and medium-term effects of both interventions in relation to the study variables to be measured. The investigators hypothesize that those patients who receive neuromodulation combined with the neuromuscular exercise program will have greater improvements.

DETAILED DESCRIPTION:
The lateral ankle complex sprain is the most prevalent musculoskeletal injury among the general population and athletes and is associated with long-term pain, disability, and high health costs. A review of ankle injuries on 70 analyzed sports established that lateral ankle sprains accounted for 77% of all injuries, where the highest incidence rates were found in sports characterized by running, changes of direction or running. jump like basketball, soccer or volleyball.One of the complications of lateral ankle sprain is the development of chronic ankle instability (CAI) characterized by repeated episodes or perceptions of ankle instability, persistent symptoms such as pain, swelling, and decreased function with limitations in activities of daily living and sports participation that persist more than a year after the initial injury. Conservative treatment is the initial therapeutic option for patients with CAI, however, the best strategies are not yet clear. Numerous rehabilitation protocols to improve CAI-associated deficits have been examined. These range from simple progressive strength work or postural dynamic balance protocols to multi-component (strength, balance, mobility) rehabilitation approaches with effective results in improving strength. , balance and in function.Clinically, a new invasive technique has appeared, known as echoguided Percutaneous Neuromodulation (EPNM). This minimally invasive intervention consists of the application of percutaneous electrical stimulation (biphasic square wave electrical current) through an acupuncture needle, as an electrode located in the vicinity of the nerve or motor point of the muscle to be treated under the guidance ultrasound where the generation of structural and excitation changes in the nerve is hypothesized, which as a consequence produces a decrease in its sensitization. It is an accessible, safe and economical technique to treat musculoskeletal conditions by physiotherapists. To date, there is limited evidence regarding its use. EPNM has been applied to different pathologies with good therapeutic results, but its use together with the combination of a multicomponent neuromuscular exercise program has never been studied.The main objective of the study will be to compare the effects in the short and medium term of an intervention with EPNM in the common peroneal nerve together with an exercise program in relation to the variables pain, range of motion in the ankle, strength of the ankle musculature , dynamic balance and functionality both in performance and in self-reports in patients with CAI.

Participants:

Voluntary subjects and adults, from the group of students of the Gimbernat University School with a history of ankle sprain and physically active, defined as participation in moderate aerobic physical activity of at least 30 minutes 5 days a week, or vigorous aerobic intensity of at least 20 minutes 3 days a week, will be evaluated to see if they can participate and be included in the study.

Variables under study:

Principal:

Self-administered scales: FAAM and CAIT. NPRS scale.

Secondaries:

Side hop test. Countermovement jump test. Star excursion balance test. Range of motion. Ankle Strength.

Randomization:

After the initial evaluation, the patients will be randomly assigned to receive a neuromuscular exercise program (control group) or to receive a neuromuscular exercise program plus a EPNM of the common peroneal nerve (experimental group). The hidden estimate is performed using a computer generated random table of numbers created prior to data collection by an outside researcher. Individualized and sequentially numbered index cards will be prepared. These will be placed in sealed opaque envelopes and the second external investigator will open the envelope and proceed with the treatment according to the screen.

Each group will be treated by a clinical physiotherapist, who will be the main investigator of the study, with more than 15 years of experience in the management of lower limb musculoskeletal injuries and more than 10 years of experience in the management of invasive techniques and ultrasound evaluation.

The researcher in charge of processing the data will be blinded with respect to belonging to the groups and likewise the researchers who will carry out the assessments will be blinded with respect to the group display of the participant. Participants in this study will not be blinded to their assigned group. All participants will read and sign an informed consent prior to inclusion in the study and will be asked to lead a lifestyle identical to the one they led before the start of the study.

Procedures:

Neuromuscular exercise program:

The strength program includes a protocol for using Theraband ® according to that described by Kaminsky et al. Participants will sit on the floor with one end of the Theraband attached to a back protector and the other end attached around the metatarsal heads of the foot to be worked on. The knee will be in full extension and the Theraband will initially be stretched to 70% of its resting length, without taking resistance into account. Strength exercises with bands will include ankle movements (dorsiflexion, inversion and eversion). The progression of the program will include an increase in series (1-3 sets of 8-10 repetitions) and an increase in resistance each week of the intervention depending on the subject's symptoms. Plantar flexion will be performed through the standing heel raise exercise. To progress the exercise in the three weeks, body weight will be taken into account. Therefore, during the first week the exercise will be performed with 30-35% of body weight, the second week with 40-45% and the third week with 50-55%.

The balance exercise program will consist of performing a series of exercises in a closed kinetic chain in a standing weight-bearing position that will be progressed from bilateral to unilateral depending on the acceptance of the load. The exercises applied in the study will be the bilateral squat and the unilateral squat in single-leg support with the maximum possible range of motion. To take into account the progress throughout the three weeks, in the bilateral squat during the first week you will work with 25-30% of the body weight, during the second week with 35-40% of the body weight and during the last week with 45-50% of body weight. In the unilateral squat you will work with 40% of the weight used in the squat each week. 3 sets of 10 repetitions will be performed.In the second week, the unilateral squat series will be performed through a backward lunge on an unstable platform (foam mat). Finally, in the third week, again with respect to the backward lunge, a disturbance will be carried out by placing a resistance band on the ankle that will favor greater activation of the muscles and in the last session a maximum range work will be carried out using assistance with a suspension system (TRX) with a weight that implies a high effort in the scale of perceived effort (8-10 points). All of these exercises will focus on motor control of the ankle, which will increase the strength of the intrinsic muscles and adequately contribute to the stabilization of the joint.

Echoguided percutaneous neuromodulation (EPNM):

The experimental group, apart from the exercise program, will receive a session of EPNM in the common peroneal nerve of the affected lower extremity. The EPNM will be applied prior to the exercise program session. 3 interventions will be carried out, in a dosage of 1 per week. It will be done with the electrostimulator (ES-160 co.).The participant will be placed in a prone position with the foot outside the stretcher. The motor part of the common peroneal nerve that affects the innervation of the superficial peroneal nerve will be searched through an Ultrasound scanner with a high-frequency linear transducer (10 Hz). A dry puncture needle (0.25mmx0.40mm, Barcelona, Spain) will be inserted until it is close to the perineurium and a biphasic symmetric square wave electric current will be applied to the needle, with a frequency of 3 Hz, a width of pulse of 250 μsec and a maximum tolerable intensity, in order to cause visible muscle contraction, according to the protocol of other studies. Ten stimulations will be performed with a duration of 10 seconds, with a rest period of 10 seconds between each stimulation. The needle will remain stationary throughout the intervention and the skin will be previously cleaned with isopropyl alcohol and chlorhexidine.

Assessment and monitoring:

The variables under study will be evaluated at 3 different times: pre-intervention measurement, post-intervention (a week after the intervention), medium-term measurement (a month after the intervention).

Adverse effects:

All patients will be asked to report any type of adverse effect they may experience throughout the study and up to one month after completion. An adverse effect is defined as a medium-term sequelae with any symptom perceived as painful or unacceptable by the participant and requiring treatment. As the introduction of the needle in some patients may induce post-treatment discomfort, subjects will be notified to report any incident. The EPNM has adverse effects that are infrequent and not serious, such as post-puncture pain that usually lasts from a few hours to a few days of mild intensity, the possible appearance of a bruise that will be minimized thanks to the use of the ultrasound and with pressure techniques on the area, the irritation of the nerve that will be minimized by the use of the ultrasound again and finally the possibility of infection, for this reason a disinfectant will be used on the area before the technique and gloves of a only use.

The therapeutic exercise program has been subsequently used by other research groups and is very safe because it is an incremental program individually adapted in intensity to each subject. Potential adverse effects are also rare, where the most common may be increased ankle pain, which will be controlled with load adaptation, possible generation of late-onset muscle soreness, which usually has a peak duration of 48 hours and a possible fall with the work of instability and disturbance, which is minimized with the presence of the therapist controlling the session at all times.

Sample size calculation:

The sample size and power calculation were calculated using the G-Power 3.1.9.4 software (Heinrich Heine Düsseldorf University).The calculations have been based using an a priori analysis with a mixed F-Anova test for repeated measures, with a Cohen's d of 0.25, a 5% level of significance (α= 0.05), 80% statistical power, two groups and 3 repeated measures(64). The estimated sample size was at least 28 subjects, 14 for each group. A dropout rate of 5% was considered during follow-up, so 15 subjects were finally included per group.

Statistical analysis of data:

1. Descriptive data in mean, range and standard deviation.
2. Normal distribution/homoscedasticity of the data (See whether the data are parametric or non-parametric).
3. Mixed-model repeated measures analysis of variance ( ANOVA) will used to see the interaction between time-group in the different variables.
4. Calculate the effect size of the difference between pre and post on the different variables with the cohen's d calculation. A effect size less than 0.2 will be considered trivial, between 0.2-0.5 low, between 0.5-0.8 moderate and greater than 0.8 high.

ELIGIBILITY:
Inclusion Criteria:

1. History of at least one major ankle sprain. The initial sprain must have occurred at least 12 months prior to study participation, be associated with inflammatory symptoms (pain, edema) and have generated at least one day of interruption in physical activity.
2. The most recent sprain must have occurred at least 3 months prior to study participation.
3. History in the injured ankle of "dropping the ankle" (at least 2 episodes in the 6 months prior to study participation) and/or repeated sprains (two or more sprains in the same ankle) and/or feelings of instability in activities of daily living or sports (score less than 24 on the Cumberland Ankle Instability Tool (CAIT).
4. Have a score of less than 75% in three or more categories in the Foot and ankle Outcome Score(FAOS) or a level of less than 80% in sports activities in the Foot and ankle ability measure (FAAM).
5. Pain on the Numeric pain rating scale (NPRS) above 3 points out of 10 in their physical activity.

Exclusion Criteria:

1. History of surgery in either of the two lower extremities that may interfere with the performance of the tests.
2. History of a fracture in either of the two lower extremities requiring alignment.
3. Acute injury to the musculoskeletal structures of other lower extremity joints in the previous 3 months, which impact joint integrity and function, resulting in at least one day of loss of physical activity.
4. Chronic concomitant pathology at the level of the lower extremity (for example: osteoarthritis, vascular disease, neural pathology).
5. Regular use of analgesic medication that may mask symptoms.
6. Contraindications of percutaneous puncture and specific to the execution of neuromodulation.
7. Being receiving physiotherapy or medical treatment during the intervention.
8. Being pregnant at the start of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
"Foot and ankle ability measure" : FAAM questionnaire | Through study completion, an average of 1 year
  It is a Likert scale that consists of 29 items, which have a score from 0 to 4, representing different levels of difficulty, divided into two subscales: activities of daily living (ADL) (21 items) and sports (8 items). items). The values are added to calculate the result of each subscale, 84 points for ADLs and 32 points for sports. For the analysis of the result, the percentage of each subscale is used separately. The test-retest reliability is high, 0.89 for the ADLs and 0.87 for the sports subscale. In fact, the FAAM scale has been shown to be valid for use in patients with ankle instability. It has been suggested that the minimal clinically important difference (MCID) is 8 and 9 points for the ADL subscale and the sports subscale, respectively.
"Cumberland Ankle Instability Tool" (CAIT) | Though study completion, an average of 1 year
  It has shown to be a valid and reliable tool to assess functional ankle instability. With an intraclass correlation coefficient (ICC) of 0.96, the CAIT scale has demonstrated excellent test-retest reliability. The scale consists of 9 items with a maximum score of 30 points, where the highest results indicate greater stability. It has been suggested that the MCID is 3 or more points.
"Numeric Pain Rating Scale" (NPRS) | Through study completion, an average of 1 year
  Scale used to assess pain intensity, where 0 is absence of pain and 10 represents maximum pain.There are no data for the MCID in patients with CAI, however it appears that changes between 1.5 and 2.1 points can be considered as the MCID for patients with musculoskeletal pain conditions. This variable will ask about the intensity of pain during sports practice.

SECONDARY OUTCOMES:
"Side hop test" (SHT) | Though study completion, an average of 1 year
  Subjects will be asked to jump laterally and medially between two tape marks that are 30 centimeters apart 10 times as fast as possible. One repetition is considered a lateral jump of 30 cm and return to the starting position. Two series will be carried out and the total time in seconds necessary to complete each of them will be recorded. Time will be recorded by a hand chronometer [ICC 0.84, Standard error measurement(SEM) 2.10 seconds and MDC 5.82 seconds]. The rest between series will be one minute and the lowest time will be used for the study. If a participant falls, puts the contralateral foot on the ground or does not correctly complete the distance of 30 cm between the lines, we consider it invalid and the participant should repeat the test.
"Countermovement jump unilateral test" (Unilateral CMJ) | Though study completion, an average of 1 year
  For this test, subjects will be asked to perform a vertical jump in a standing position with their hands placed on their pelvis. To do this, there will first be a descent phase where the subjects will flex the knee approximately 90 degrees to then take off as quickly as possible keeping the lower extremity extended during the flight phase. The extremity that we do not value will remain at all times without contact on the ground. There will be 3 repetitions with a 30-second rest between each one where we will stay with the highest value. For the measurement, the My Jump 2 application will be used. The validity of the application has been seen to be high (ICC= 0.997, 95% (Intraclass Coefficient (CI): 0.996-0.998, P < 0.001) with an almost perfect correlation coefficient (r= 0.995, P< 0.001) between the application and the gold standard, which is a force platform.
Isometric ankle strength measurement | Though study completion, an average of 1 year
  Measurement of three muscle groups: the inverters, the evertors/plantarflexors, the inverters/dorsiflexors. Isometric assessment of the ankle in inversion/dorsiflexion and in eversion/plantarflexion selectively assesses the tibialis anterior and peroneus longus and brevis muscles, respectively. The measurement will be made with the Microfet2 hand pressure dynamometer (Hogan Scientific, LLC, Salt Lake City, USA. (ICC 0.61, 95% CI=0.09-0.81 for dorsiflexors, ICC 0.74, 95% CI= 0.425-0.879 for inverters and ICC 0.84, 95% CI=0.431-0.905 for evertors in the standardized positions to ensure consistency throughout the study. For this variable, 3 measurements of 5 seconds duration will be carried out with 20 seconds of rest between measurements. The value to take into account will be the peak isometric force in kg and will be normalized with the body mass of the subjects.
"Star Excursion Balance Test" (SEBT) | Though study completion, an average of 1 year
  Is a measure of dynamic balance that has been shown to be valid with moderate to good reliability.The 3 SEBT directions to be measured are the anterior, the posterolateral and the posteromedial, as support to previous investigations (ICC intra 0.85-0.91 and ICC inter 0.99-1) with reported minimum detectable change values (MDC). ) of the normalized reach distance of 5.9% for the anterior direction, 7.8% for the posteromedial direction, and 7.6% for the posterolateral direction. 3 consecutive measurements will be made in each direction. The order of the addresses will be randomized.
Range of Motion (ROM) | Though study completion, an average of 1 year
  Ankle dorsiflexion range of motion will be measured with the My Rom app (version 3.0.4). Its validity has been demonstrated with respect to the Limit® mini digital inclinometer (r = 0.989, 95% CI = 0.986-0.993) and its reliability (ICC = 0.976, 95% CI = 0.966- 0.983, Dorsiflex app Coefficient of variation(CV) = 5.1 ± 2.3%; Digital inclinometer CV = 4.9 ± 2.5%) during the lunge test under load.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Ortega, Study Director — Universidad Rey Juan Carlos
Locations (1):
- Escuelas Universitarias Gimbernat, Torrelavega, Cantabria, Spain

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data

REFERENCES:
- [Background] Fernandez-de-Las-Penas C, Ortega-Santiago R, De-la-Llave-Rincon AI, Cleland JA, Pareja JA, Fahandezh-Saddi-Diaz H, Arias-Buria JL. Ultrasound-guided percutaneous electrical nerve stimulation versus surgery for women with unilateral carpal tunnel syndrome: A randomized parallel-group trial. Eur J Pain. 2023 Aug;27(7):860-870. doi: 10.1002/ejp.2117. Epub 2023 Apr 7. PMID 36987682
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Carlesso LC, Macdermid JC, Santaguida LP. Standardization of adverse event terminology and reporting in orthopaedic physical therapy: application to the cervical spine. J Orthop Sports Phys Ther. 2010 Aug;40(8):455-63. doi: 10.2519/jospt.2010.3229. PMID 20710083
- [Background] David P, Halimi M, Mora I, Doutrellot PL, Petitjean M. Isokinetic testing of evertor and invertor muscles in patients with chronic ankle instability. J Appl Biomech. 2013 Dec;29(6):696-704. doi: 10.1123/jab.29.6.696. Epub 2013 Jan 18. PMID 23343782
- [Background] Kim KJ, Kim YE, Jun HJ, Lee JS, Ji SH, Ji SG, Seo TH, Kim YO. Which Treatment is More Effective for Functional Ankle Instability: Strengthening or Combined Muscle Strengthening and Proprioceptive Exercises? J Phys Ther Sci. 2014 Mar;26(3):385-8. doi: 10.1589/jpts.26.385. Epub 2014 Mar 25. PMID 24707089
- [Background] Balsalobre-Fernandez C, Romero-Franco N, Jimenez-Reyes P. Concurrent validity and reliability of an iPhone app for the measurement of ankle dorsiflexion and inter-limb asymmetries. J Sports Sci. 2019 Feb;37(3):249-253. doi: 10.1080/02640414.2018.1494908. Epub 2018 Jul 2. PMID 29962280
- [Background] Salaffi F, Stancati A, Silvestri CA, Ciapetti A, Grassi W. Minimal clinically important changes in chronic musculoskeletal pain intensity measured on a numerical rating scale. Eur J Pain. 2004 Aug;8(4):283-91. doi: 10.1016/j.ejpain.2003.09.004. PMID 15207508
- [Background] Kendrick DB, Strout TD. The minimum clinically significant difference in patient-assigned numeric scores for pain. Am J Emerg Med. 2005 Nov;23(7):828-32. doi: 10.1016/j.ajem.2005.07.009. PMID 16291435
- [Background] Jensen MP, Turner JA, Romano JM, Fisher LD. Comparative reliability and validity of chronic pain intensity measures. Pain. 1999 Nov;83(2):157-62. doi: 10.1016/s0304-3959(99)00101-3. PMID 10534586
- [Background] Collins CK, Masaracchio M, Cleland JA. The effectiveness of strain counterstrain in the treatment of patients with chronic ankle instability: A randomized clinical trial. J Man Manip Ther. 2014 Aug;22(3):119-28. doi: 10.1179/2042618614Y.0000000069. PMID 25125933
- [Background] Alfuth M, Hahm MM. RELIABILITY, COMPARABILITY, AND VALIDITY OF FOOT INVERSION AND EVERSION STRENGTH MEASUREMENTS USING A HAND-HELD DYNAMOMETER. Int J Sports Phys Ther. 2016 Feb;11(1):72-84. PMID 26900502
- [Background] Mentiplay BF, Perraton LG, Bower KJ, Adair B, Pua YH, Williams GP, McGaw R, Clark RA. Assessment of Lower Limb Muscle Strength and Power Using Hand-Held and Fixed Dynamometry: A Reliability and Validity Study. PLoS One. 2015 Oct 28;10(10):e0140822. doi: 10.1371/journal.pone.0140822. eCollection 2015. PMID 26509265
- [Background] Bogataj S, Pajek M, Hadzic V, Andrasic S, Padulo J, Trajkovic N. Validity, Reliability, and Usefulness of My Jump 2 App for Measuring Vertical Jump in Primary School Children. Int J Environ Res Public Health. 2020 May 25;17(10):3708. doi: 10.3390/ijerph17103708. PMID 32466091
- [Background] Caffrey E, Docherty CL, Schrader J, Klossner J. The ability of 4 single-limb hopping tests to detect functional performance deficits in individuals with functional ankle instability. J Orthop Sports Phys Ther. 2009 Nov;39(11):799-806. doi: 10.2519/jospt.2009.3042. PMID 19881005
- [Background] Wright CJ, Linens SW, Cain MS. Establishing the Minimal Clinical Important Difference and Minimal Detectable Change for the Cumberland Ankle Instability Tool. Arch Phys Med Rehabil. 2017 Sep;98(9):1806-1811. doi: 10.1016/j.apmr.2017.01.003. Epub 2017 Jan 27. PMID 28137476
- [Background] Hiller CE, Refshauge KM, Bundy AC, Herbert RD, Kilbreath SL. The Cumberland ankle instability tool: a report of validity and reliability testing. Arch Phys Med Rehabil. 2006 Sep;87(9):1235-41. doi: 10.1016/j.apmr.2006.05.022. PMID 16935061
- [Background] Cruz-Diaz D, Hita-Contreras F, Lomas-Vega R, Osuna-Perez MC, Martinez-Amat A. Cross-cultural adaptation and validation of the Spanish version of the Cumberland Ankle Instability Tool (CAIT): an instrument to assess unilateral chronic ankle instability. Clin Rheumatol. 2013 Jan;32(1):91-8. doi: 10.1007/s10067-012-2095-0. Epub 2012 Oct 9. PMID 23053687
- [Background] Eechaute C, Vaes P, Van Aerschot L, Asman S, Duquet W. The clinimetric qualities of patient-assessed instruments for measuring chronic ankle instability: a systematic review. BMC Musculoskelet Disord. 2007 Jan 18;8:6. doi: 10.1186/1471-2474-8-6. PMID 17233912
- [Background] Martin RL, Irrgang JJ, Burdett RG, Conti SF, Van Swearingen JM. Evidence of validity for the Foot and Ankle Ability Measure (FAAM). Foot Ankle Int. 2005 Nov;26(11):968-83. doi: 10.1177/107110070502601113. PMID 16309613
- [Background] Cervera-Garvi P, Ortega-Avila AB, Morales-Asencio JM, Cervera-Marin JA, Martin RR, Gijon-Nogueron G. Cross-cultural adaptation and validation of Spanish version of The Foot and Ankle Ability Measures (FAAM-Sp). J Foot Ankle Res. 2017 Aug 22;10:39. doi: 10.1186/s13047-017-0221-6. eCollection 2017. PMID 28852426
- [Background] Haskell WL, Lee IM, Pate RR, Powell KE, Blair SN, Franklin BA, Macera CA, Heath GW, Thompson PD, Bauman A. Physical activity and public health: updated recommendation for adults from the American College of Sports Medicine and the American Heart Association. Med Sci Sports Exerc. 2007 Aug;39(8):1423-34. doi: 10.1249/mss.0b013e3180616b27. PMID 17762377
- [Background] de la Cruz-Torres B, Barrera-Garcia-Martin I, Albornoz-Cabello M. Immediate effects of ultrasound-guided percutaneous neuromodulation versus physical exercise on performance of the flexor hallucis longus muscle in professional dancers: a randomised clinical trial. Acupunct Med. 2019 Apr;37(2):91-97. doi: 10.1177/0964528419826103. Epub 2019 Mar 12. PMID 30860393
- [Background] De-la-Cruz-Torres B, Carrasco-Iglesias C, Minaya-Munoz F, Romero-Morales C. Crossover effects of ultrasound-guided percutaneous neuromodulation on contralateral hamstring flexibility. Acupunct Med. 2021 Oct;39(5):512-521. doi: 10.1177/0964528420920283. Epub 2020 May 13. PMID 32403999
- [Background] Terada M, Harkey MS, Wells AM, Pietrosimone BG, Gribble PA. The influence of ankle dorsiflexion and self-reported patient outcomes on dynamic postural control in participants with chronic ankle instability. Gait Posture. 2014;40(1):193-7. doi: 10.1016/j.gaitpost.2014.03.186. Epub 2014 Apr 3. PMID 24768526
- [Background] Hall EA, Chomistek AK, Kingma JJ, Docherty CL. Balance- and Strength-Training Protocols to Improve Chronic Ankle Instability Deficits, Part I: Assessing Clinical Outcome Measures. J Athl Train. 2018 Jun;53(6):568-577. doi: 10.4085/1062-6050-385-16. Epub 2018 Jul 5. PMID 29975573
- [Background] Sekir U, Yildiz Y, Hazneci B, Ors F, Aydin T. Effect of isokinetic training on strength, functionality and proprioception in athletes with functional ankle instability. Knee Surg Sports Traumatol Arthrosc. 2007 May;15(5):654-64. doi: 10.1007/s00167-006-0108-8. Epub 2006 Jun 13. PMID 16770637
- [Background] Mettler A, Chinn L, Saliba SA, McKeon PO, Hertel J. Balance training and center-of-pressure location in participants with chronic ankle instability. J Athl Train. 2015 Apr;50(4):343-9. doi: 10.4085/1062-6050-49.3.94. Epub 2015 Jan 6. PMID 25562457
- [Background] Mattacola CG, Lloyd JW. Effects of a 6-week strength and proprioception training program on measures of dynamic balance: a single-case design. J Athl Train. 1997 Apr;32(2):127-35. PMID 16558442
- [Background] Hale SA, Hertel J, Olmsted-Kramer LC. The effect of a 4-week comprehensive rehabilitation program on postural control and lower extremity function in individuals with chronic ankle instability. J Orthop Sports Phys Ther. 2007 Jun;37(6):303-11. doi: 10.2519/jospt.2007.2322. PMID 17612356
- [Background] Eils E, Rosenbaum D. A multi-station proprioceptive exercise program in patients with ankle instability. Med Sci Sports Exerc. 2001 Dec;33(12):1991-8. doi: 10.1097/00005768-200112000-00003. PMID 11740289
- [Background] McKeon PO, Ingersoll CD, Kerrigan DC, Saliba E, Bennett BC, Hertel J. Balance training improves function and postural control in those with chronic ankle instability. Med Sci Sports Exerc. 2008 Oct;40(10):1810-9. doi: 10.1249/MSS.0b013e31817e0f92. PMID 18799992
- [Background] Wright CJ, Linens SW, Cain MS. A Randomized Controlled Trial Comparing Rehabilitation Efficacy in Chronic Ankle Instability. J Sport Rehabil. 2017 Jul;26(4):238-249. doi: 10.1123/jsr.2015-0189. Epub 2016 Aug 24. PMID 27632874
- [Background] Linens SW, Ross SE, Arnold BL. Wobble Board Rehabilitation for Improving Balance in Ankles With Chronic Instability. Clin J Sport Med. 2016 Jan;26(1):76-82. doi: 10.1097/JSM.0000000000000191. PMID 25831410
- [Background] Kidgell DJ, Horvath DM, Jackson BM, Seymour PJ. Effect of six weeks of dura disc and mini-trampoline balance training on postural sway in athletes with functional ankle instability. J Strength Cond Res. 2007 May;21(2):466-9. doi: 10.1519/R-18945.1. PMID 17530947
- [Background] Smith BI, Docherty CL, Simon J, Klossner J, Schrader J. Ankle strength and force sense after a progressive, 6-week strength-training program in people with functional ankle instability. J Athl Train. 2012 May-Jun;47(3):282-8. doi: 10.4085/1062-6050-47.3.06. PMID 22892409
- [Background] Kaminski TW, Buckley BD, Powers ME, Hubbard TJ, Ortiz C. Effect of strength and proprioception training on eversion to inversion strength ratios in subjects with unilateral functional ankle instability. Br J Sports Med. 2003;37(5):410-5; discussion 415. doi: 10.1136/bjsm.37.5.410. PMID 14514531
- [Background] Hall EA, Docherty CL, Simon J, Kingma JJ, Klossner JC. Strength-training protocols to improve deficits in participants with chronic ankle instability: a randomized controlled trial. J Athl Train. 2015 Jan;50(1):36-44. doi: 10.4085/1062-6050-49.3.71. Epub 2014 Nov 3. PMID 25365134
- [Background] Docherty CL, Moore JH, Arnold BL. Effects of strength training on strength development and joint position sense in functionally unstable ankles. J Athl Train. 1998 Oct;33(4):310-4. PMID 16558526
- [Background] Goulart Neto AM, Maffulli N, Migliorini F, de Menezes FS, Okubo R. Validation of Foot and Ankle Ability Measure (FAAM) and the Foot and Ankle Outcome Score (FAOS) in individuals with chronic ankle instability: a cross-sectional observational study. J Orthop Surg Res. 2022 Jan 21;17(1):38. doi: 10.1186/s13018-022-02925-9. PMID 35062990
- [Background] Baczkowicz D, Falkowski K, Majorczyk E. Assessment of Relationships Between Joint Motion Quality and Postural Control in Patients With Chronic Ankle Joint Instability. J Orthop Sports Phys Ther. 2017 Aug;47(8):570-577. doi: 10.2519/jospt.2017.6836. Epub 2016 Nov 4. PMID 27814667
- [Background] Zhang L, Lu J, Cai B, Fan S, Jiang X. Quantitative assessments of static and dynamic balance performance in patients with chronic ankle instability. Medicine (Baltimore). 2020 Apr;99(17):e19775. doi: 10.1097/MD.0000000000019775. PMID 32332619
- [Background] Kosik KB, Johnson NF, Terada M, Thomas AC, Mattacola CG, Gribble PA. Decreased dynamic balance and dorsiflexion range of motion in young and middle-aged adults with chronic ankle instability. J Sci Med Sport. 2019 Sep;22(9):976-980. doi: 10.1016/j.jsams.2019.05.005. Epub 2019 May 10. PMID 31122877
- [Background] Pollock AS, Durward BR, Rowe PJ, Paul JP. What is balance? Clin Rehabil. 2000 Aug;14(4):402-6. doi: 10.1191/0269215500cr342oa. PMID 10945424
- [Background] Gribble PA, Hertel J, Denegar CR, Buckley WE. The Effects of Fatigue and Chronic Ankle Instability on Dynamic Postural Control. J Athl Train. 2004 Dec;39(4):321-329. PMID 15592604
- [Background] Hoch MC, Staton GS, Medina McKeon JM, Mattacola CG, McKeon PO. Dorsiflexion and dynamic postural control deficits are present in those with chronic ankle instability. J Sci Med Sport. 2012 Nov;15(6):574-9. doi: 10.1016/j.jsams.2012.02.009. Epub 2012 May 8. PMID 22575498
- [Background] Wisthoff B, Matheny S, Struminger A, Gustavsen G, Glutting J, Swanik C, Kaminski TW. Ankle Strength Deficits in a Cohort of College Athletes With Chronic Ankle Instability. J Sport Rehabil. 2019 Sep 1;28(7):752-757. doi: 10.1123/jsr.2018-0092. PMID 30222475
- [Background] Donnelly L, Donovan L, Hart JM, Hertel J. Eversion Strength and Surface Electromyography Measures With and Without Chronic Ankle Instability Measured in 2 Positions. Foot Ankle Int. 2017 Jul;38(7):769-778. doi: 10.1177/1071100717701231. Epub 2017 Apr 9. PMID 28391722
- [Background] Al Adal S, Pourkazemi F, Mackey M, Hiller CE. The Prevalence of Pain in People With Chronic Ankle Instability: A Systematic Review. J Athl Train. 2019 Jun;54(6):662-670. doi: 10.4085/1062-6050-531-17. Epub 2019 Jun 11. PMID 31184959
- [Background] Hershkovich O, Tenenbaum S, Gordon B, Bruck N, Thein R, Derazne E, Tzur D, Shamiss A, Afek A. A large-scale study on epidemiology and risk factors for chronic ankle instability in young adults. J Foot Ankle Surg. 2015 Mar-Apr;54(2):183-7. doi: 10.1053/j.jfas.2014.06.001. Epub 2014 Aug 16. PMID 25135102
- [Background] Martin RL, Davenport TE, Paulseth S, Wukich DK, Godges JJ; Orthopaedic Section American Physical Therapy Association. Ankle stability and movement coordination impairments: ankle ligament sprains. J Orthop Sports Phys Ther. 2013 Sep;43(9):A1-40. doi: 10.2519/jospt.2013.0305. No abstract available. PMID 24313720
- [Background] Tanen L, Docherty CL, Van Der Pol B, Simon J, Schrader J. Prevalence of chronic ankle instability in high school and division I athletes. Foot Ankle Spec. 2014 Feb;7(1):37-44. doi: 10.1177/1938640013509670. Epub 2013 Nov 27. PMID 24287210
- [Background] Lin CI, Houtenbos S, Lu YH, Mayer F, Wippert PM. The epidemiology of chronic ankle instability with perceived ankle instability- a systematic review. J Foot Ankle Res. 2021 May 28;14(1):41. doi: 10.1186/s13047-021-00480-w. PMID 34049565
- [Background] Arnold BL, Wright CJ, Ross SE. Functional ankle instability and health-related quality of life. J Athl Train. 2011 Nov-Dec;46(6):634-41. doi: 10.4085/1062-6050-46.6.634. PMID 22488189
- [Background] Hertel J, Corbett RO. An Updated Model of Chronic Ankle Instability. J Athl Train. 2019 Jun;54(6):572-588. doi: 10.4085/1062-6050-344-18. Epub 2019 Jun 4. PMID 31162943
- [Background] Gribble PA, Delahunt E, Bleakley C, Caulfield B, Docherty CL, Fourchet F, Fong D, Hertel J, Hiller C, Kaminski TW, McKeon PO, Refshauge KM, van der Wees P, Vicenzino B, Wikstrom EA. Selection criteria for patients with chronic ankle instability in controlled research: a position statement of the International Ankle Consortium. J Orthop Sports Phys Ther. 2013 Aug;43(8):585-91. doi: 10.2519/jospt.2013.0303. Epub 2013 Jul 31. PMID 23902805
- [Background] Fong DT, Hong Y, Chan LK, Yung PS, Chan KM. A systematic review on ankle injury and ankle sprain in sports. Sports Med. 2007;37(1):73-94. doi: 10.2165/00007256-200737010-00006. PMID 17190537
- [Background] Gribble PA, Bleakley CM, Caulfield BM, Docherty CL, Fourchet F, Fong DT, Hertel J, Hiller CE, Kaminski TW, McKeon PO, Refshauge KM, Verhagen EA, Vicenzino BT, Wikstrom EA, Delahunt E. 2016 consensus statement of the International Ankle Consortium: prevalence, impact and long-term consequences of lateral ankle sprains. Br J Sports Med. 2016 Dec;50(24):1493-1495. doi: 10.1136/bjsports-2016-096188. Epub 2016 Jun 3. PMID 27259750
- [Background] Gribble PA, Bleakley CM, Caulfield BM, Docherty CL, Fourchet F, Fong DT, Hertel J, Hiller CE, Kaminski TW, McKeon PO, Refshauge KM, Verhagen EA, Vicenzino BT, Wikstrom EA, Delahunt E. Evidence review for the 2016 International Ankle Consortium consensus statement on the prevalence, impact and long-term consequences of lateral ankle sprains. Br J Sports Med. 2016 Dec;50(24):1496-1505. doi: 10.1136/bjsports-2016-096189. Epub 2016 Jun 3. PMID 27259753

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/17/NCT05942417/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/17/NCT05942417/ICF_001.pdf